CLINICAL TRIAL: NCT01481506
Title: Efficacy Of Multiparametric Telemonitoring On Respiratory Outcomes In Elderly People With Chronic Obstructive Pulmonary Disease.
Brief Title: Multiparametric Telemonitoring In Elderly People With Chronic Obstructive Pulmonary Disease
Acronym: SweetAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Raffaele Antonelli Incalzi, Director, Unit of Geriatrics., Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 29/2009 ComEt CBM - SweetAge
Record Dates: First submitted 2011-11-08; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemonitoring (Experimental)
  Interventions: Procedure: Telemonitoring
- Usual care (No Intervention)

INTERVENTIONS:
Procedure: Telemonitoring — Use of wearable sensors for heart rate, haemoglobin oxygen saturation, physical activity, respiratory rate with automatic transmission to the monitoring central.
  Arms: Telemonitoring

SUMMARY:
Chronic obstructive pulmonary disease (COPD) determines an important risk of disability and disease-related need of care. Selected interventions were able to reduce the number and the severity of exacerbations. Telemedicine has also been proposed for this purpose. Current evidences, however, are scant. The investigators present a randomized, parallel-group trial of a multiparametric remote monitoring system to test its ability to improve early exacerbation detection rates and impact on clinical outcomes.

DETAILED DESCRIPTION:
All patients performed a simple spirometry that was carried out using a Stead-Wells bell spirometer (Biomedin, Padua, Italy). Upon provision of informed consent, patients in the telemonitoring group were invited to a session during which they were instructed on how to wear the wristband and to operate the cellular telephone. A study physician was available on call during office hours to assist patients needing further instructions. A technician was also available in order to solve ingoing hardware problems.

All participants were also clinically evaluated at baseline and received a multi-dimensional assessment including: Activities of daily living scale (ADL), Instrumental activities of daily living scale (IADL), Mini-mental state examination (MMSE) test. These are well validated and routinely used tools to screen geriatric patients in order to detect global, physical and instrumental autonomy and consequent degree of dependence, as well as cognitive status.

Patients in both groups were followed up for 9 months, during this period they attended the standard schedule of clinical controls. For patients in the SweetAge group, the parameters received were evaluated daily by a study physician. In case of abnormal readings, the physician systematically contacted the patient to verify whether their symptoms had worsened or new symptoms had arose. In this event, the patient's adherence to her/his therapy was checked and, if unsatisfactory, individually tailored interventions promoting adherence were carried up. Otherwise, a diagnosis of exacerbation was made and, on the basis of its severity, an outpatient clinical assessment (for mild exacerbations) or a hospital admission was scheduled.

The outcome measures of these study were: number of exacerbations (defined as a sustained worsening of the patient's condition, from the stable state and beyond normal day-to-day variations, that is acute in onset and necessitates a change in regular medications, and number of hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic obstructive pulmonary disease stage II-III (GOLD classification)

Exclusion Criteria:

* Cognitive impairment precluding the use of the experimental device.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Respiratory Events | 9 months
  Rate of COPD exacerbations, defined as a sustained worsening of the patient's condition, from the stable state and beyond normal day-to-day variations, that is acute in onset and necessitates a change in regular medications. Rate of hospital admission for respiratory problems (COPD exacerbations, lower respiratory tract infections, respiratory failure).

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, MD, Principal Investigator — Campus BioMedico University

REFERENCES:
- [Derived] Pedone C, Chiurco D, Scarlata S, Incalzi RA. Efficacy of multiparametric telemonitoring on respiratory outcomes in elderly people with COPD: a randomized controlled trial. BMC Health Serv Res. 2013 Mar 6;13:82. doi: 10.1186/1472-6963-13-82. PMID 23497109